CLINICAL TRIAL: NCT03836820
Title: Effects of Clinical Pilates Exercises in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Songul Baglan Yentur, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 436
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arhritis; Pilates exercises; Fatigue
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinical pilates exercise (Experimental): Clinical pilates exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Interventions: Other: Clinical pilates exercise; Other: Clinical Pilates and Aerobic Exercise
- Aerobic exercise (Experimental): Progressive aerobic walking exercise will be performed three days in a week. Exercise intensity will be 50- 80% of maximal heart rate and exercises will be performed 45 minutes in per session for 8 weeks.
  Interventions: Other: Aerobic exercise; Other: Clinical Pilates and Aerobic Exercise
- Clinical pilates and Aerobic exercise (Experimental): Both clinical pilates exercises and progressive aerobic walking exercises will be performed three days in a week for 8 weeks.
  Interventions: Other: Clinical pilates exercise; Other: Aerobic exercise; Other: Clinical Pilates and Aerobic Exercise

INTERVENTIONS:
Other: Clinical pilates exercise — Clinical pilates exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Arms: Clinical pilates and Aerobic exercise; Clinical pilates exercise
Other: Aerobic exercise — Progressive aerobic walking exercise will be performed three days in a week. Exercise intensity will be 50- 80% of maximal heart rate and exercises will be performed 45 minutes in per session for 8 weeks.
  Arms: Aerobic exercise; Clinical pilates and Aerobic exercise
Other: Clinical Pilates and Aerobic Exercise — Both clinical pilates exercises and progressive aerobic walking exercises will be performed three days in a week for 8 weeks.

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease characterised by polyarthritis and erosive synovitis. Articular and extraarticular sympthoms are mostly seen in patients with RA. Additionally, extra complaints such as depression, fatigue, kinesiophobia and physical inactivity may accompany. Positive effects of physical activity and exercise are known. In some studies, effects of pilates exercises have been investigated on many different diseases such as Multiple Sclerosis, Ankylosing Spondylitis and breast cancer. The aim of this study is to investigate effects of clinical pilates exercises on fatigue, depression, aerobic capacity, pain, quality of life, disease activity and sleep quality.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease characterised by polyarthritis and erosive synovitis and is associated with progressive impairments and activity limitations. It may cause destruction of bone and cartilage by affecting synovial joints symmetrically. Organ involvement may be seen in the patients with RA as well as joint involvement. Initiation of the disease is mostly insidious and varies from patient to patient. Hand, wrist, foot, elbow and knee joints involvement are common. Furthermore almost all joints may be affected. Extraarticular symptoms are subcutaneous nodules, visceral nodules, cardiologic involvement, pulmonary involvement, eye involvement, neurological involvement, vasculitis, felty syndrome, amyloidosis, osteoporosis, liver and renal involvements. These symptoms may cause some extra complaints such as depression, fatigue, kinesiophobia and physical inactivity. Studies in literature have reported reduction in physical activity level in patients with RA. Reasons of physical inactivity can be listed as general obstacles such as lack of time, lack of motivation, weather condition and disease related blocks such as pain, fatigue, disease activity, depression, kinesiophobia. Depression prevalence in RA patients is found between 14.8% and 38.8% and this rate is estimated five times more than healthy people. Also, a study investigating pain in RA patients resulted that pain may be correlated with fatigue and depression. Fatigue which is frequently observed complaint of patients with rheumatic diseases is reported incidence between 40% and 80%. RA patients have been reported at high risk for cardiovascular diseases in EULAR recommendations.

Positive effects of physical activity and exercise on physiological, morphological and psychosocial conditions are known. Endurance, flexibility, muscle strength, body composition, self confidence and mood improve by regular exercise and high physical activity level. Furthermore, anti-inflammatory affects of exercise are proved in last years. Aims of pilates exercises which are developed by Joseph Pilates are to increase motor control, range of motion, flexibility, muscle strength and endurance, to improve balance, respiratory pattern and body awareness, to reduce stress. There are many studies investigating affects of pilates exercises on quality of life, functional capacity, posture, pain for different diseases including Multiple Sclerosis, Ankylosing Spondylitis, breast cancer. Aerobic and strengthening exercises reported to have positive affects on fatigue, quality of life, depression and pain for RA patients. The aim of this study is to investigate effects of clinical pilates exercises on fatigue, depression, aerobic capacity, pain, quality of life, disease activity and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 to 65 and who have diagnosed with RA according to American College of Rheumatology criteria will be included the study.

Exclusion Criteria:

* Patients who were pregnant, diagnosed with malignancy, had changes of medical treatment in the last 3 months, had dysfunction that limited physical activity such as severe neurological impairment, immobility or cooperation deficits, had regular exercise habit (minimally three days in a week), had high disease activity score (DAS-28>3.2) and had cardiac symphtoms according to New YorkHeart Association will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-24 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity | 6 minutes
  The 6-minute walk test is a submaximal exercise test used to quantify the functional exercise capacity in clinical populations. It measures the distance walked within a period of 6-minutes.
Fatigue severity scale | 2 minutes
  Fatigue is a normal response to physical exertion or stress but can also be a sign of a physical disorder. In the common sense, fatigue is a condition known to everyone from his or her own experience,irrespective of his or her age, gender, or health. Fatigue severity scale consists of nine questions; each question is scored from 1 to 7

SECONDARY OUTCOMES:
Beck Depression Inventory | 2 minutes
  The Beck Depression Inventory (BDI) is world-wide among the most used selfrating scales for measuring depression. BDI consists of 21 items related to depressive symptoms such as pessimism, sense of failure, guilt, dissatisfaction, sleep, appetite and fatigue. Each item is scored between 0 and 3. Total score is 63, and an increase of the score means increased severity of depression. According to this scale 1-10 points are defined as normal, scores between 11-16 indicate mild mental distress, 17-20 indicate the patient is at the border points for clinical depression, 21-30 indicate moderate depression, severe depression scores are between 31-40 and 40 points above are interpreted as a very serious depression.
Short Form McGill Pain Questionnaire | 1 minute
  This questionnaire consists of 11 sensory and 4 affective descriptive words. These 15 words are described as 0 = absent, 1 = mild, 2 = moderate, 3 = severe pain. So three type of pain scores (sensory, affective, total = sensory + affective) are obtained. In McGill Pain Questionnaire, the current level of pain is measured by Visual Analog Scale (VAS) and Likert scale consisting of 6 points (0 = no pain, 1 = mild, 2 = irritating, 3 = bothersome, 4 = terrible, 5 = unbearable).
Pittsburgh Sleep Quality | 2 minutes
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.
Disease Activity Score- 28 | 10 minutes
  Disease Activity Score (DAS) is an assessment tool used to measure the level of disease activity in patients with RA. The DAS combines information from swollen joints, tender joints, erythrocyte sedimentation rate (ESR), and patient self-report of general health
The Rheumatoid Arthritis Quality of Life Questionnaire | 2 minutes
  The Rheumatoid Arthritis Quality of Life (RAQoL) questionnaire is a disease-specific quality of life measure that was developed simultaneously in the UK and the Netherlands. The content of the RAQoL was derived from in-depth qualitative interviews with RA patients exploring.
  the impact of RA on their QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Deran Oskay, Study Director — Gazi University Faculty of Health Sciences
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Munsterman T, Takken T, Wittink H. Are persons with rheumatoid arthritis deconditioned? A review of physical activity and aerobic capacity. BMC Musculoskelet Disord. 2012 Oct 18;13:202. doi: 10.1186/1471-2474-13-202. PMID 23078261
- [Result] Rongen-van Dartel SA, Repping-Wuts H, Flendrie M, Bleijenberg G, Metsios GS, van den Hout WB, van den Ende CH, Neuberger G, Reid A, van Riel PL, Fransen J. Effect of Aerobic Exercise Training on Fatigue in Rheumatoid Arthritis: A Meta-Analysis. Arthritis Care Res (Hoboken). 2015 Aug;67(8):1054-62. doi: 10.1002/acr.22561. PMID 25624016
- [Derived] Yentur SB, Atas N, Ozturk MA, Oskay D. Comparison of the effectiveness of pilates exercises, aerobic exercises, and pilates with aerobic exercises in patients with rheumatoid arthritis. Ir J Med Sci. 2021 Aug;190(3):1027-1034. doi: 10.1007/s11845-020-02412-2. Epub 2020 Oct 22. PMID 33094465